CLINICAL TRIAL: NCT05266625
Title: Randomized, Controlled, Multicenter, Pragmatic, Trial With Open-label Extension of BT-001 to Improve Glycemic Control in Adults With Type 2 Diabetes in a Real-world Setting
Brief Title: Digital Therapeutic Based Investigation to Improve Glycemic Control in Patients With Type 2 Diabetes and Residual Hyperglycemia on Stable Medical Therapy
Acronym: BRIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Better Therapeutics (Industry)
Collaborators: CPC Clinical Research (Unknown); University of Colorado, Denver (Other); Ascension Health (Industry); Department of Veterans Affairs Hospital Durham, NC (Unknown); University of Colorado Health Clinics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM2-07-CPC
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to an intervention arm or control arm. After 6 months, patients in the control arm will be able to cross over to using the intervention.
Masking Description: While patients and providers will not be told which arm they are in, it will be obvious when they complete the installation of the mobile application which arm they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention BT-001 + Standard of Care (Experimental): Patients in this arm will receive the BT-001 treatment for up to 720 days.
  Interventions: Behavioral: BT-001
- Standard of Care (Other): Patients will have access to a control mobile application for 180 days and then will have the option to use the treatment for the remainder of the 720 day study
  Interventions: Other: Control App

INTERVENTIONS:
Behavioral: BT-001 — Bt-001 is a software application that delivers treatment to participants with type 2 diabetes, using behavioral therapy. BT-001 is accessed via the participants' smartphone.
  The behavioral intervention process involves:
  Identifying maladaptive thoughts based on misinformed core beliefs that lead to disease-promoting behaviors; replacing maladaptive core beliefs with adaptive ways of thinking; and providing collaborative construction of behavioral exercises to test core beliefs.
  Each week, Bt-001 asks participants to complete a new lesson, along with one skill exercise. The lessons are expected to take between 10-20 minutes to complete. In addition to completing a lesson and skill, participants will be directed to report plant-based meals consumed and minutes of exercise completed and to measure their blood sugar daily.
  Arms: Intervention BT-001 + Standard of Care
Other: Control App — The app asks patients brief questions about their health but does not include any behavioral therapy.
  Arms: Standard of Care

SUMMARY:
Randomized, controlled, multicenter, pragmatic, pivotal trial with open-label extension evaluating the hypothesis that BT-001 an investigational digital therapeutic intended to help patients with type 2 diabetes improve their glycemic control, will lower hemoglobin A1c (HbA1c) compared to a control application added to usual care and across a broad range of patients in a real-world setting

DETAILED DESCRIPTION:
This randomized, controlled, multicenter, parallel-arm, pragmatic pivotal trial with extension will evaluate the hypothesis that BT-001 compared to a control application, both on top of usual care, will lower HbA1c in real world clinical practice. Approximately five-hundred (500) adults with type 2 diabetes will be randomized (1:1) to BT-001 or the control application. Most clinical data will be collected via the electronic medical records (EMR) system with limited additional contacts to ascertain adverse device effects (ADEs), adverse events (AEs) and clinical events which may have occurred outside the health system and were not recorded in the EMR. For primary efficacy endpoint assessment, a requisition form for HbA1c at a local laboratory will be provided if HbA1c is not available from the EMR within the 90- and 180-day time windows. During the extension phase, biomarker endpoint data will only be collected from the EMR. For all participants, clinical and healthcare utilization data will be extracted from their EMR for the period from 180 days prior to enrollment to 720 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, inclusive at the time of signing the informed consent
* Type 2 diabetes on stable anti-diabetic regimen for at least three (3) months
* HbA1c 7.0% to 10.9% (within thirty [30] days of signing the informed consent form [ICF])
* Able to use BT-001 e.g., English fluent, smartphone is capable of running the study intervention.

Exclusion Criteria:

* Current use of outpatient prandial insulin
* In the opinion of the investigator, life expectancy < one (1) year
* COVID-19 diagnosis within thirty (30) days prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 90 days
  Difference in the mean change from baseline in HbA1c between treatment groups.
Adverse Events | 90 days
  Occurrence, relatedness and severity of adverse device effects and adverse events between treatment groups

SECONDARY OUTCOMES:
Difference in HbA1c | 180 days
  Difference in mean change from baseline in HbA1c between treatment groups.
Adverse Events | 180 days
  Occurrence, relatedness and severity of adverse device effects and adverse events between treatment groups

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - Ascension DePaul Community Health, New Orleans, Louisiana
  - VA Medical Center-Durham, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD